CLINICAL TRIAL: NCT05359705
Title: Comparison of Motion and Comfort for Thoracolumbosacral Orthoses - Group 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: More Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4051
Record Dates: First submitted 2022-01-13; First posted 2022-05-04 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Back Injuries
MeSH Terms: conditions — Back Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): Healthy subjects who meet the Inclusion/Exclusion.
  Interventions: Device: DJO 456; Device: Aspen 456; Device: DJO 464; Device: Aspen 464

INTERVENTIONS:
Device: DJO 456 — Data will be recorded while subjects wear a 456 back brace manufactured by DJO Global
Device: Aspen 456 — Data will be recorded while subjects wear a 456 back brace manufactured by Aspen Medical Products
Device: DJO 464 — Data will be recorded while subjects wear a 464 back brace manufactured by DJO Global
Device: Aspen 464 — Data will be recorded while subjects wear a 464 back brace manufactured by Aspen Medical Products

SUMMARY:
The study will measure and compare range of motion (ROM), motion during simulated activities of daily living ADL), tissue interface pressure (TIP), muscle activation (EMG), and trunk stiffness and damping measurements (TSD) for two pairs of back braces: Postural TLSO (456), and TLSO (464).

ELIGIBILITY:
Inclusion Criteria:

* BMI < 40
* English speaking
* Subjects who have read and signed IRB approved informed consent for this study
* Of appropriate body size for back brace per instructions for use

Exclusion Criteria:

* History of back pain or back injury requiring medical care within the previous 12 months
* History of spinal surgery, physical or chiropractic therapy of the back
* History of spinal spondylosis or osteoporosis
* Pregnant
* Currently Incarcerated

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
Flexion - Sagittal plane | Day 1
  Angle of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects flex their trunk relative to their pelvis in the sagittal plane.
Extension - Sagittal plane | Day 1
  Angle of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects extend their trunk relative to their pelvis in the sagittal plane.
Range of motion - Frontal plane | Day 1
  Range of motion of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects bend their trunk relative to their pelvis laterally to the right and left in the frontal plane.
Range of motion - Transverse plane | Day 1
  Range of motion of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects rotate their trunk relative to their pelvis laterally to the right and left in the transverse plane.
Rotation angle while looking over shoulder | Day 1
  Maximum rotation angle of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects rotate their trunk relative to their pelvis to look at an object placed 150 degrees behind them.
Range of motion in the sagittal plane when rising from a chair | Day 1
  Range of motion in the sagittal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects rise from a chair.
Range of motion in the sagittal plane when returning to a seated position | Day 1
  Range of motion in the sagittal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects move from an upright standing position to a seated position.
Flexion angle in the sagittal plane when touching right hallux in a seated position | Day 1
  Range of motion in the sagittal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach forward and down to touch their right hallux while in a seated position.
Flexion angle in the sagittal plane when picking an object up from the floor | Day 1
  Range of motion in the sagittal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach forward and down to pick up a 85mm diameter object weighing 500grams from the floor from a standing position.
Range of motion in the sagittal plane while walking on a level surface | Day 1
  Range of motion in the sagittal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects walk across a level surface.
Range of motion in the frontal plane while walking on a level surface | Day 1
  Range of motion in the frontal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects walk across a level surface.
Range of motion in the transverse plane while walking on a level surface | Day 1
  Range of motion in the transverse plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects walk across a level surface.
Range of motion in the sagittal plane while ascending stairs. | Day 1
  Range of motion in the sagittal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects ascend a flight of four steps
Range of motion in the sagittal plane while descending stairs. | Day 1
  Range of motion in the sagittal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects descend a flight of four steps
Range of motion in the frontal plane while ascending stairs. | Day 1
  Range of motion in the frontal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects ascend a flight of four steps
Range of motion in the frontal plane while descending stairs. | Day 1
  Range of motion in the frontal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects descend a flight of four steps
Range of motion in the transverse plane while ascending stairs. | Day 1
  Range of motion in the transverse plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects ascend a flight of four steps
Range of motion in the transverse plane while descending stairs. | Day 1
  Range of motion in the transverse plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects descend a flight of four steps
Flexion angle in the sagittal plane when reaching forwards and around an object with their right hand. | Day 1
  Flexion angle in the sagittal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach forwards and around the back of a chair with their right hand
Flexion angle in the sagittal plane when reaching forwards and around an object with their left hand. | Day 1
  Flexion angle in the sagittal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach forwards and around the back of a chair with their left hand
Lateral angle in the frontal plane when reaching forwards and around an object with their right hand. | Day 1
  Lateral angle in the frontal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach forwards and around the back of a chair with their right hand
Lateral angle in the frontal plane when reaching forwards and around an object with their left hand. | Day 1
  Lateral angle in the frontal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach forwards and around the back of a chair with their left hand
Rotation angle in the transverse plane when reaching forwards and around an object with their right hand. | Day 1
  Rotation angle in the transverse plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach forwards and around the back of a chair with their right hand
Rotation angle in the transverse plane when reaching forwards and around an object with their left hand. | Day 1
  Rotation angle in the transverse plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach forwards and around the back of a chair with their left hand
Flexion angle in the sagittal plane when reaching when reach down to pick up a suitcase | Day 1
  Flexion angle in the sagittal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach down to pick up a standard carry-on sized suitcase positioned to the right of their body with their right hand
Lateral angle in the frontal plane when reaching when reach down to pick up a suitcase | Day 1
  Lateral angle in the frontal plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach down to pick up a standard carry-on sized suitcase positioned to the right of their body with their right hand
Rotation angle in the transverse plane when reaching when reach down to pick up a suitcase | Day 1
  Rotation angle in the transverse plane of the thorax relative to the pelvis will be measured in degrees using stereophotogrammetric techniques while subjects reach down to pick up a standard carry-on sized suitcase positioned to the right of their body with their right hand

SECONDARY OUTCOMES:
Comfort | Day 1
  Subjects will be asked to provide a subjective rating of brace comfort using a 10cm visual analog comfort rating scale for each of the back braces during all ROM and ADL testing conditions. The endpoints of the scale will be labeled "Very comfortable", and "Very uncomfortable" at 0 and 10cm respectively.
Trunk stiffness and damping - front angle | Day 1
  Each subject will kneel in a apparatus with their pelvis fixed in position and their trunk upright. A load will be attached to front of their upper body and a force applied. The force will be released and subsequent upper trunk motion measured using an inertial measurement unit. Maximum angular motion of the upper body in degrees will be measured.
Trunk stiffness and damping - front angular velocity | Day 1
  Each subject will kneel in a apparatus with their pelvis fixed in position and their trunk upright. A load will be attached to front of their upper body and a force applied. The force will be released and subsequent upper trunk motion measured using an inertial measurement unit. Maximum angular velocity of the upper body after force release will be measured in degrees/second.
Trunk stiffness and damping - front angular acceleration | Day 1
  Each subject will kneel in a apparatus with their pelvis fixed in position and their trunk upright. A load will be attached to front of their upper body and a force applied. The force will be released and subsequent upper trunk motion measured using an inertial measurement unit. Maximum angular acceleration of the upper body after force release will be measured in degrees/second/second.
Trunk stiffness and damping - back angle | Day 1
  Each subject will kneel in a apparatus with their pelvis fixed in position and their trunk upright. A load will be attached to back of their upper body and a force applied. The force will be released and subsequent upper trunk motion measured using an inertial measurement unit. Maximum angular motion of the upper body in degrees will be measured.
Trunk stiffness and damping - back angular velocity | Day 1
  Each subject will kneel in a apparatus with their pelvis fixed in position and their trunk upright. A load will be attached to back of their upper body and a force applied. The force will be released and subsequent upper trunk motion measured using an inertial measurement unit. Maximum angular velocity of the upper body after force release will be measured in degrees/second.
Trunk stiffness and damping - back angular acceleration | Day 1
  Each subject will kneel in a apparatus with their pelvis fixed in position and their trunk upright. A load will be attached to back of their upper body and a force applied. The force will be released and subsequent upper trunk motion measured using an inertial measurement unit. Maximum angular acceleration of the upper body after force release will be measured in degrees/second/second.
Trunk stiffness and damping - right side angle | Day 1
  Each subject will kneel in a apparatus with their pelvis fixed in position and their trunk upright. A load will be attached to right side of their upper body and a force applied. The force will be released and subsequent upper trunk motion measured using an inertial measurement unit. Maximum angular motion of the upper body in degrees will be measured.
Trunk stiffness and damping - right side angular velocity | Day 1
  Each subject will kneel in a apparatus with their pelvis fixed in position and their trunk upright. A load will be attached to right side of their upper body and a force applied. The force will be released and subsequent upper trunk motion measured using an inertial measurement unit. Maximum angular velocity of the upper body after force release will be measured in degrees/second.
Trunk stiffness and damping - right side angular acceleration | Day 1
  Each subject will kneel in a apparatus with their pelvis fixed in position and their trunk upright. A load will be attached to right side of their upper body and a force applied. The force will be released and subsequent upper trunk motion measured using an inertial measurement unit. Maximum angular velocity of the upper body after force release will be measured in degrees/second/second.

OTHER OUTCOMES:
Left Iliocostalis muscle activity (AUC) - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left iliocostalis muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Left Iliocostalis muscle activity (AUC) - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left iliocostalis muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Right Iliocostalis muscle activity (AUC) - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right iliocostalis muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Right Iliocostalis muscle activity (AUC) - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right iliocostalis muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Maximum left Iliocostalis muscle activity - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left iliocostalis muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum left Iliocostalis muscle activity - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left iliocostalis muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum right Iliocostalis muscle activity - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right iliocostalis muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum right Iliocostalis muscle activity - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right iliocostalis muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Left longissimus muscle activity (AUC) - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left Longissimus muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Left longissimus muscle activity (AUC) - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left Longissimus muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Right longissimus muscle activity (AUC) - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right Longissimus muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Right longissimus muscle activity (AUC) - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right Longissimus muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Maximum left longissimus muscle activity - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left Longissimus muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum left longissimus muscle activity - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left Longissimus muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum right longissimus muscle activity - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right Longissimus muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum right longissimus muscle activity - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right Longissimus muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Left external oblique muscle activity (AUC) - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left external oblique muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Left external oblique muscle activity (AUC) - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left external oblique muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Right external oblique muscle activity (AUC) - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right external oblique muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Right external oblique muscle activity (AUC) - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right external oblique muscle. After filtering the muscle signal, the average area under the curve during one gait cycle will be calculated and reported for each back brace as a percentage for the area under the curve when subjects were not wearing a back brace.
Maximum left external oblique muscle activity - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left external oblique muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum left external oblique muscle activity - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the left external oblique muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum right external oblique muscle activity - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right external oblique muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum right external oblique muscle activity - stair ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right external oblique muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Right rectus abdominus muscle activity (AUC) - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right rectus abdominus muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Right rectus abdominus muscle activity (AUC) - stair aseent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right rectus abdominus muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum right rectus abdominus muscle activity - walking | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right rectus abdominus muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.
Maximum right rectus abdominus muscle activity - ascent | Day 1
  A low profile surface electrode will be used to record the electromyographic activity of the right rectus abdominus muscle. After filtering the muscle signal, the maximum value during one gait cycle will be calculated and reported for each back brace as a percentage for the maximum value when subjects were not wearing a back brace.

CONTACTS AND LOCATIONS:
Locations (1):
- MORE Foundation, Phoenix, Arizona, United States